CLINICAL TRIAL: NCT05982652
Title: Heart Rate Variability and Its Association With Symptom of Orthostatic Hypotension in Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Hae-ri Park, doctor, Pusan National University Yangsan Hospital
Other Study IDs: 05-2021-293
Record Dates: First submitted 2022-10-13; First posted 2023-08-08 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Spinal Cord Injuries; Orthostatic Hypotension; Heart Rate Variability
Keywords: Spinal Cord Injuries; Orthostatic Hypotension; Heart rate variability; Autonomic nervous system
MeSH Terms: conditions — Spinal Cord Injuries; Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-OH group: without orthostaric hypotension in spinal cord injuries
- symptomatic OH group: Symptomatic individuals in a patient population diagnosed with orthostatic hypotension (Symptom : dizziness, visual disturbance, nausea and headache)
- asymptomatic OH group: Asymptomatic individuals in a patient population diagnosed with orthostatic hypotension

SUMMARY:
In this study, the SCI patients were sub-grouped on the basis of symptoms into symptomatic and asymptomatic groups and measured HRV during resting and tilt up tests to compare their cardiovascular autonomic functions.

DETAILED DESCRIPTION:
In study protocol and the subjects were asked to lie down quietly for 5 minutes, closing their eyes and avoiding talking, moving hand, legs and body, and coughing during the test. R-R interval and blood pressure were measured beat-to-beat using Finometer® PRO (Finapres Medical Systems, Amsterdam, Netherlands) for 6 minutes each in two positions, supine and 60-degree angle on the tilt table.

ELIGIBILITY:
Inclusion Criteria:

* spinal cord injury with or without OH
* aged 19 or older
* ASIA Impairment Scale (AIS) A to D
* neurological level of injury above T6.

Exclusion Criteria:

* Those with heart and respiratory diseases, neurological diseases other than SCI - medically unstable states
* Those who are taking medications affecting BP that cannot be stopped

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with SCI were recruited from a single university-affiliated rehabilitation hospital.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences of heart rate variability between groups (OH vs non-OH, asymptomatic-OH vs symptomatic-OH group) | at the test time (15minutes)
  mean HR (heart rate), mean RR(RR interval), RMSSD (mean square of the successive R-R interval differences), SDNN (standard deviation of normal-to-normal interval), LF (low frequency) domain, HF(High frequency) domain
Logistic regression analysis of heart rate variability variables according to OH and presence of symptom | at the test time (15minutes)
  the investigators conducted logistic regression analysis to evaluate the significance and impact of HRV variables associated with orthostatic hypotension and its symptoms in spinal cord injury patients.

CONTACTS AND LOCATIONS:
Overall Officials: PARK HAERI, Master, Study Director — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Geumo-ro 20, Mulgeum-eup, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stampas A, Zhu L, Li S. Heart rate variability in spinal cord injury: Asymptomatic orthostatic hypotension is a confounding variable. Neurosci Lett. 2019 Jun 11;703:213-218. doi: 10.1016/j.neulet.2019.03.020. Epub 2019 Mar 20. PMID 30904574